CLINICAL TRIAL: NCT00227994
Title: Donepezil/ Galantamine in the Treatment of Post-stroke Cognitively Impaired Rehabilitating Elderly
Brief Title: Acetylcholinesterase Inhibitors to Improve Cognitive Function and Overall Rehabilitation After a Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Eric Lenze, Professor of Psychiatry, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23MH064196-01 (NIH); K23MH064196-01 (NIH)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Cerebrovascular Accident
Keywords: Cholinesterase Inhibitors; Elderly; Stroke; Cognition
MeSH Terms: conditions — Stroke | interventions — Galantamine; Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Galantamine (Experimental): Galantamine for 12 weeks
  Interventions: Drug: Galantamine
- Donepezil (Experimental): Donepezil for 12 weeks
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Galantamine — Participants assigned to receive galantamine will receive 4 mg twice a day for 4 weeks, 8 mg twice a day for the next 4 weeks, and 12 mg twice a day for the remainder of the study.
  Other Names: Razadyne
  Arms: Galantamine
Drug: Donepezil — Participants assigned to receive donepezil will receive 5 mg twice a day for 6 weeks, and then 10 mg twice a day for the next 6 weeks.
  Other Names: Aricept
  Arms: Donepezil

SUMMARY:
This study will evaluate the effectiveness of treatment with acetylcholinesterase inhibitors in improving cognitive function and overall rehabilitation in elderly stroke survivors.

DETAILED DESCRIPTION:
Cognitive impairment is a common result of a stroke and can be detrimental to recovery. It can negatively affect both mental and physical functioning, thereby complicating the rehabilitation process. Although much research has targeted the effects of long-term cognitive impairment after a stroke, very little research has been done to examine the incidence and course of cognitive impairment during the first three months following a stroke. These first three months are the most important in terms of regaining function. Acetylcholinesterase inhibitors have been beneficial to both sufferers of vascular dementia and Alzheimer's disease. They may also be a useful pharmacologic intervention to enhance post-stroke rehabilitation. This study will compare the effectiveness of two acetylcholinesterase inhibitors, galantamine and donepezil, in improving cognitive function and overall rehabilitation in elderly stroke survivors.

Participants in this open label study will be randomly assigned to receive either galantamine or donepezil for 12 weeks. Participants assigned to receive galantamine will receive 4 mg twice a day for 4 weeks, 8 mg twice a day for the next 4 weeks, and 12 mg twice a day for the remainder of the study. Participants assigned to receive donepezil will receive 5 mg twice a day for 6 weeks, and then 10 mg twice a day for the next 6 weeks. Functional independence will be measured at baseline and Weeks 2 and 12. In addition, a pre-stroke level of functional independence will be obtained through a structured interview with participants and their families. Participants will also be monitored for signs of depression and medication side effects throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a rehabilitation hospital with primary diagnosis of ischemic stroke (cardiovascular accident)
* Stroke was within 30 days of being admitted
* Medically stable
* Presence of memory and/or attentional impairments and evidence that these impairments were not present or were less severe prior to the stroke (assessed via interview with family)
* Approval by individual's attending physician at the rehabilitation hospital

Exclusion Criteria:

* Aphasia or cognitive (or behavioral) impairments severe enough to prevent valid neuropsychiatric assessment
* Currently experiencing a major depressive episode (unless treated and in partial remission, assessed using the Primary Care Evaluation of Mental Disorders)
* Current psychosis or mania
* History of substance or alcohol abuse or dependence within three months of study entry
* Currently taking a cholinomimetic drug
* Medical condition with known sensitivity to donepezil (e.g., slower than normal heart rate, supraventricular cardiac conduction defects, severe asthma or obstructive pulmonary disease, active upper gastrointestinal bleed, or gastric/duodenal ulcer if not on acid-blocking agent)
* Informed that taking donepezil is medically inadvisable
* Current use of any anticholinergic medication (e.g., for bladder spasm)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-04; Primary Completion 2005-01 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Lenze, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
study has small sample size and is unlikely to be useful for data sharing efforts; however, interested researchers can contact the first author via email.

REFERENCES:
- [Result] Whyte EM, Lenze EJ, Butters M, Skidmore E, Koenig K, Dew MA, Penrod L, Mulsant BH, Pollock BG, Cabacungan L, Reynolds CF 3rd, Munin MC. An open-label pilot study of acetylcholinesterase inhibitors to promote functional recovery in elderly cognitively impaired stroke patients. Cerebrovasc Dis. 2008;26(3):317-21. doi: 10.1159/000149580. Epub 2008 Jul 31. PMID 18667813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 participants received study medication
Period: Overall Study
Arm/Group | Galantamine | Donepezil
Started | 20 | 20
Completed | 13 | 13
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galantamine | Donepezil | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (7.5) | 69.1 (6.4) | 69.5 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Physical Function (Measured by the FIM-motor)
Description: Score on Functional Independence Measure (FIM) motor score, where 7 indicates total assistance/complete dependence and 91 is complete independence
Time Frame: Measured at weeks 0 and 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine | Donepezil
Number analyzed (Participants) | 13 | 13
units on a scale
  Baseline FIM | 47.1 (9.7) | 49.4 (8.34)
  Week 12 FIM | 73.1 (16.5) | 87.4 (5.2)

2. Secondary Outcome: Medication Tolerability
Description: Number of participants who withdrew due to side effects.
Time Frame: Measured throughout the study
Measure: Number; unit: participants
Arm/Group | Galantamine | Donepezil
Number analyzed (Participants) | 20 | 20
participants | 5 | 5

ADVERSE EVENTS:
Arm/Group | Galantamine | Donepezil
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less